CLINICAL TRIAL: NCT05001412
Title: Clinical Study of Chemotherapy Combined With Camrelizumab and Apatinib in First-line Treatment of Extensive Stage Small Cell Lung Cancer
Brief Title: Chemotherapy Combined With Camrelizumab and Apatinib in First-line Treatment of ES-SCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhou Chengzhi (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Zhou Chengzhi, Professor, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CROC-2021
Record Dates: First submitted 2021-07-22; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: Camrelizumab; apatinib
MeSH Terms: interventions — camrelizumab; apatinib; Carboplatin; Etoposide

STUDY DESIGN:
Intervention Model Description: We divide them into two cohorts based on the extent of tumor invasion to the mediastinum or hilar large vessels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort one (Experimental): Extensive SCLC patients who are Peripheral type or tumor vascular invasion grade one or less.
  Interventions: Drug: Camrelizumab; apatinib; carboplatin; etoposide
- Cohort two (Experimental): Extensive SCLC patients who are central type or tumor vascular invasion grade two to three.
  Interventions: Drug: Camrelizumab; apatinib; carboplatin; etoposide

INTERVENTIONS:
Drug: Camrelizumab; apatinib; carboplatin; etoposide — 2 cycle chemotherapy (carboplatin and etoposide), and then 2 cycle chemotherapy (carboplatin and etoposide) combine with Camrelizumab and apatinib, finally maintenance therapy with Camrelizumab and apatinib

SUMMARY:
The efficacy of PD-1/PD-L1 combined with chemotherapy in the treatment of extensive small-cell lung cancer is still unsatisfactory. PD-1/PD-L1 combined with chemotherapy and anti-angiogenic drugs may achieve better efficacy.

DETAILED DESCRIPTION:
Camrelizumab is a humanized PD-1 monoclonal antibody. Camrelizumab combined with the antiangiogenic drug apatinib has achieved good efficacy in extensive small-cell lung cancer. Median OS is 8.4 months. In our study, subjects with extensive stage small cell lung cancers receive 2 cycles of chemotherapy followed by carrizumab combined with apatinib and chemotherapy. we hope to achieve a better outcome.

ELIGIBILITY:
Inclusion Criteria:

* 1. Extensive stage small cell lung cancer proved by pathology.
* 2. Extensive small cell lung cancer does not receive systematic treatment.
* 3. limited SCLC patients have received radiotherapy and chemotherapy for more than 6 months.
* 4. patients have measurable lesions according to RECIST version 1.1.
* 5. Male or female who is 18 to 75 years old.
* 6. ECOG PS 0 or 1.
* 7. Life expectancy is more than12 weeks.
* 8. Appropriate organ system function.
* 9. hyroid-stimulating hormone is ULN or less (If T3 and T4 is normal, he still meets the Inclusion Criteria even the abnormal TSH. )
* 10. Take proper contraceptive measures.
* 11. Subjects voluntarily participate in this study and sign the informed consent.

Exclusion Criteria:

* 1. Previous treatment with apatinib, anti-programmed cell death (PD-1), anti-PD-1, or other PD-1/ PD-L1 immunotherapy.
* 2. Cancer meningitis.
* 3. patients had been diagnosed and/or treated for other malignancies within 5 years prior to enrollment, except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix.
* 4. There are many factors affecting oral medication, such as inability to swallow, post-gastrointestinal resection, chronic diarrhea, intestinal obstruction, etc..
* 5. Uncontrollable pleural effusion, pericardial effusion or ascites, requiring repeated drainage.
* 6. Patients with spinal cord compression who were not cured or relieved by surgery and/or radiotherapy, or who were diagnosed with spinal cord compression after treatment and without clinical evidence of stable disease ≥1 week before enrollment;
* 7. Patients with hypertension who cannot be well controlled by oral antihypertensive therapy, suffer from myocardial ischemia or myocardial infarction of grade I or above, arrhythmias of grade I or above , or cardiac insufficiency;
* 8. Subjects had signs of bleeding, hemoptysis, or a history of unhealed wounds, ulcers, fractures within 2 months prior to initial administration.
* 9. The adverse events caused by previous treatment did not completely recover.
* 10. Patients with major surgery or obvious traumatic injury within 28 days before enrollment;
* 11. Occurred arterial or venous thromboembolism events within 6 months.
* 12. People with a history of drug abuse or mental disorders.
* 13. Suffering from a serious and/or uncontrollable disease;
* 14. Vaccination or attenuated vaccine received within 4 weeks.
* 15. Severe allergies that require treatment with other monoclonal antibody drugs;
* 16. Active autoimmune disease requiring systemic treatment within 2 years prior to the first administration;
* 17. Immunosuppressive therapy with systemic or absorbable local hormones and continued for 2 weeks after the first dose;
* 18. Participate in other anticancer drug clinical trials within 4 weeks;
* 19. In the investigator's judgment, there are other factors that may have led to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-01-25 (Estimated); Study Completion 2024-01-25 (Estimated)

PRIMARY OUTCOMES:
Safety: Dose-limiting toxicities | Followed up every 3 weeks.
  Any level 4 or greater hematologic toxicity and any level 3 or greater non-hematologic toxicity (accroding to CTC AE 5.0)

SECONDARY OUTCOMES:
PFS | Imageological diagnosis every 6 weeks
  Progression Free Survival
12 months OS | Followed up by telephone every 2 months
  12 months overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Chengzhi Zhou, MD, Study Director — The First Affiliated Hospital of Guangzhou Medical University; Xin Chen, MD, Principal Investigator — Zhujiang Hospital affiliated to Southern Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
No plan.

REFERENCES:
- [Derived] Liu M, Qiu G, Guan W, Xie X, Lin X, Xie Z, Zhang J, Qin Y, Du H, Chen X, Deng Y, Li S, Zhong N, Zhou C. Induction chemotherapy followed by camrelizumab plus apatinib and chemotherapy as first-line treatment for extensive-stage small-cell lung cancer: a multicenter, single-arm trial. Signal Transduct Target Ther. 2025 Feb 18;10(1):65. doi: 10.1038/s41392-025-02153-7. PMID 39962074